CLINICAL TRIAL: NCT06928246
Title: Pilot Study on Cellular and Molecular Impact of Neuroimmune Interactions in Atopic Dermatitis
Brief Title: The Impact of Botox on Neuroimmune Interactions in Atopic Dermatitis
Acronym: AD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel Kaplan (Other)
Collaborators: Almirall, S.A. (Industry)
Responsible Party: Sponsor-Investigator, Daniel Kaplan, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: STUDY24110067
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Atopic dermatitis; Eczema; Botox
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Onabotulinum Toxin Type A - Phase 1b (Experimental): Onabotulinum toxin administered to two lesions.
  Interventions: Drug: Onabotulinum Toxin Type A - Phase 1b
- Onabotulinum Toxin Type A - Phase 2 (Experimental): Onabotulinum toxin administered to three lesions.
  Interventions: Drug: Onabotulinum Toxin Type A - Phase 2

INTERVENTIONS:
Drug: Onabotulinum Toxin Type A - Phase 1b — The lesions receiving Botulinum toxin will get five 0.1 mL intradermal injections of 5 units of Botulinum toxin which equates to 25 units per lesion and 50 units per patient.
  Arms: Onabotulinum Toxin Type A - Phase 1b
Drug: Onabotulinum Toxin Type A - Phase 2 — The lesions receiving Botulinum toxin will get five 0.1 mL intradermal injections of 5 units of Botulinum toxin which equates to 25 units per lesion and 75 units per patient.
  Arms: Onabotulinum Toxin Type A - Phase 2

SUMMARY:
The purpose of this study is to understand cellular and molecular interactions in the skin of participants with mild-to-moderate AD, and how botulinum toxin alters these interactions.

DETAILED DESCRIPTION:
Atopic dermatitis is a debilitating chronic inflammatory disease with substantial health and economic impact, affecting 10-20% of the U.S. population with an estimated annual direct health care cost of $13 billion. There is much to still discover regarding the dysfunctional skin barrier underlying AD and its effects on quality of life, highlighting a critical health care cap. AD manifests as erythematous and pruritic plaques often in flexural regions of the body, but may also be widespread as well. AD patients suffer from high rates of mental health disorders and often report a poor quality of life (QoL).

The pathogenesis of AD is multifactorial, involving both genetic and environmental components. Specifically, a defect in the filaggrin gene is a common etiology. Moreover, it is thought that decreased levels of ceramides within the epidermis allow for an abnormal amount of transepidermal water loss leading to an increased Th2 response and subsequently, overexpression of proinflammatory cytokines IL-4 and IL-5. Additionally, scratching of the epidermis promotes increased levels of IL-1, IL-6 and TNF-alpha from keratinocytes.

The objective of this pilot study is to determine whether cutaneous neurons are required for the maintenance of atopic dermatitis (AD) lesions. The significance derives from the potential to reveal novel neuro-immune pathways that could provide suitable targets for future therapeutic approaches for this disease. Specifically, the investigators hypothesize that neurotransmitters released from cutaneous neurons are required for the persistence of AD lesions. This is supported by a prior report showing that injection of botulinum toxin which prevents vesicular fusion in neurons and hence neurotransmitter release led to clinical improvement and resolution of AD lesions. Similar findings have been reported with Psoriasis. The investigators approach will analyze biopsy samples from AD patients treated with botulinum toxin using spatial single cell imaging.

The project will be performed in 2 phases. Phase 1a will include a pilot run of spatial single cell imaging performed on normal skin and with atopic dermatitis. In Phase 1b, the investigators will administer intradermal botulinum toxin in AD lesions to determine the kinetics of the clinical response when neurotransmitter release is inhibited using standardized clinical outcome assessments, including Physician Global Assessment (PGA) and Eczema Area and Severity Index (EASI). The kinetics, or time, to reduction of lesion severity, as determined in Phase 1b, will be used in Phase 2 to determine the biopsy visits.

Phase 2 will test the hypothesis that botulinum toxin therapy alters the cellular and molecular state of AD lesions, specifically by blocking neuroimmune interactions with a specific emphasis of cytokine and chemokine interactions. In Phase 2, botulinum toxin will be injected into multiple lesions in a small cohort of AD patients. Based on the results of Phase 1b, skin biopsies will be harvested at 3 different times and analyzed using spatial single cell imaging.

It is expected that these experiments will implicate neuroimmune interactions in the pathogenesis of AD and serve as proof-of-concept for design of randomized controlled trials (RCTs) evaluating the efficacy of botulinum toxin to reduce inflammation, lesion severity, and improve quality of life for AD patients. Once patients are clear, inhibition of neurotransmitter release could be used to prevent recurrence thereby avoiding long-term immunosuppression and its associated risks.

ELIGIBILITY:
Inclusion Criteria:

Phase 1b:

* Patients 18 years or older at time of consent
* Mild-to-Moderate AD, defined as:
* BSA ≤ 10%
* IGA ≤ 3
* No past biologic therapy
* No systemic therapy for 3 months
* No topical therapy for treatment of AD for 4 weeks

Phase 2:

* Patients 18 years or older at time of consent
* Mild-to-Moderate AD, defined as:
* BSA ≤ 10%
* IGA ≤ 3
* At least one patch of eczema of at least 5 cm in diameter
* No past biologic therapy
* No systemic therapy for 3 months
* No topical therapy for treatment of AD for 4 weeks

Exclusion Criteria:

Phase 1b:

* Age less than 18 years old
* Pregnant or breastfeeding
* Has medical comorbidity such as end stage congestive heart failure or coagulopathy that is a relative contradiction to skin biopsy procedure
* Has had prior exposure to biologic treatments or has had prior treatment with systemic non-biologics (e.g. methotrexate) within 12 weeks
* Has used topical therapy for treatment of AD within 4 weeks

Phase 2:

* Patients enrolled in Phase 1
* Age less than 18 years old
* Pregnant or breastfeeding
* Has medical comorbidity such as end stage congestive heart failure or coagulopathy that is a relative contradiction to skin biopsy procedure
* Has had prior exposure to biologic treatments or has had prior treatment with systemic non-biologics (e.g. methotrexate) within 12 weeks
* Has used topical therapy for treatment of AD within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percentage change in EASI scores at Day 28 as compared to baseline. | At Day 28
  Eczema Area and Severity Index (EASI) total score from 0-72, with higher score indicating more severity. The EASI index assigns proportionate values to 4 body regions. Each region is assigned a score of 0 to 3, indicating none, mild, moderate, and severe clinical expression. The percentage of area involved is also assigned an eruption proportional score from 0 to 6. The total body score for each body region is obtained by multiplying the sum of the severity scores by the area score, then multiplying the result by the constant weighted value assigned to that body region. The sum of these scores gives the EASI total from 0-72.
Percentage change in PGA at Day 28 as compared to baseline. | At Day 28
  The Physician's Global Assessment (PGA) is a clinician-reported measure used to assess the overall severity of atopic dermatitis (AD) at a single time point. It utilizes a scale of 5-points; total scale ranging from 0 (clear) to 5 (severe disease). The PGA score represents overall disease severity based on clinical signs including erythema, induration/papulation, lichenification, and oozing/crusting. Higher scores indicate greater disease severity.

SECONDARY OUTCOMES:
Percentage change in transcriptional mRNA in immune and non-immune cells in skin biopsies, up to Day 28, as compared to baseline. | Until last biopsy, up to Day 28
  Skin biopsies used to analyze transcriptional mRNA in immune and non-immune cells. Expression levels tested by Xenium Spatial Cell Imaging; a high-resolution, spatial transcriptomics platform used to perform single-cell resolution analysis of cell populations by mapping their gene expression profiles.
Percentage change in spatial distribution of specific cell types in skin biopsies, up to Day 28, as compared to baseline. | Until last biopsy, up until Day 28
  Skin biopsies used to analyze spatial location of immune and non-immune cells. Expression levels tested by Xenium Spatial Cell Imaging; a high-resolution, spatial transcriptomics platform used to perform single-cell resolution analysis of cell populations by mapping their spatial distribution profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kaplan, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD can be made available to researchers in a closed environment for a specified period of time.
Supporting Information: Study Protocol, CSR
Time Frame: From end of study up to two years.
Access Criteria: Data-sharing is subject to approved scientifically sound research proposal and signed data-sharing agreement.

REFERENCES:
- [Background] Popescu MN, Beiu C, Iliescu MG, Mihai MM, Popa LG, Stanescu AMA, Berteanu M. Botulinum Toxin Use for Modulating Neuroimmune Cutaneous Activity in Psoriasis. Medicina (Kaunas). 2022 Jun 16;58(6):813. doi: 10.3390/medicina58060813. PMID 35744076
- [Background] Khattab FM. Evaluation of Botulinum Toxin A as an Optional Treatment for Atopic Dermatitis. J Clin Aesthet Dermatol. 2020 Jul;13(7):32-35. Epub 2020 Jul 1. PMID 32983334